CLINICAL TRIAL: NCT07101744
Title: Iparomlimab and Tuvonralimab Combined With Nimotuzumab in Recurrent or Metastatic Nasopharyngeal Carcinoma After First-line Treatment Failure: A Single-arm Phase IIa Clinical Trial
Brief Title: Iparomlimab and Tuvonralimab Combined With Nimotuzumab in Recurrent or Metastatic NPC After First-line Treatment Failure: A Single-arm Phase IIa Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fei Han, Principal lnvestigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-381-01
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma (NPC); First-line Treatment Failure Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma (NPC); Nimotuzumab; Iparomlimab and Tuvonralimab
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental group (Experimental): Iparomlimab and Tuvonralimab combined with Nimotuzumab , administered on Day 1 every 3 weeks (D1 Q3W), until disease progression or unacceptable toxicity，or for a maximum of one year
  Interventions: Drug: Iparomlimab and Tuvonralimab

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — Iparomlimab and Tuvonralimab combined with Nimotuzumab , administered on Day 1 every 3 weeks (D1 Q3W), until disease progression or unacceptable toxicity.

SUMMARY:
This study aims to preliminarily explore the efficacy and safety of Iparomlimab and Tuvonralimab in combination with Nimotuzumab for the treatment of recurrent/metastatic nasopharyngeal carcinoma (NPC). It is expected to investigate a novel therapeutic regimen with improved efficacy and enhanced safety for recurrent/metastatic NPC, thereby providing robust evidence-based medical support for the application of dual-target immune checkpoint inhibitors in nasopharyngeal carcinoma therapy

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score of 0-1;
2. Age 18 to 70 years;
3. Histologically confirmed nasopharyngeal carcinoma;
4. Patients with locoregional recurrence unsuitable for surgery or radiotherapy, or those who developed distant metastasis after standard comprehensive treatment, or initially diagnosed with metastatic nasopharyngeal carcinoma, provided they have experienced treatment failure with first-line cisplatin-based regimens (± PD-1 monoclonal antibody);
5. Availability of nasopharyngeal + neck MRI data prior to enrollment, with at least one measurable lesion (excluding bone metastases);
6. Willingness to provide archived tumor tissue specimens or undergo a biopsy to collect tumor tissue for PD-L1 expression level testing;
7. Laboratory test results within 7 days prior to enrollment meeting the following criteria:

   Hematology: Absolute neutrophil count (ANC) ≥ 2.0 × 10^9/L, hemoglobin (Hb) ≥ 9.0 g/dL, platelets (PLT) ≥ 100 × 10^9/L;

   Liver function: Total bilirubin < 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.5 × ULN;

   Renal function: Serum creatinine < 1.5 × ULN.
8. Voluntary participation with signed informed consent form.

Exclusion Criteria:

1. History of other malignancies (except adequately treated non-melanoma skin cancer, in situ carcinoma, or other cancers cured ≥5 years prior);
2. Comorbidities requiring long-term immunosuppressive therapy or systemic/local corticosteroids at immunocompromising doses;
3. Immunodeficiency diseases or history of organ transplantation (including but not limited to: interstitial pneumonia, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.);
4. HIV-positive status; HBsAg-positive with detectable HBV DNA ≥1000 copies/mL; or HCV antibody-positive;
5. High-dose glucocorticoid use within 4 weeks prior;
6. Pregnant/lactating women or individuals of reproductive potential without effective contraception;
7. Laboratory test abnormalities beyond protocol-defined thresholds within 7 days before enrollment;
8. Significant impairment of cardiac, hepatic, pulmonary, renal, or bone marrow function;
9. Uncontrolled comorbidities or active infections;
10. Concurrent participation in other clinical trials or receipt of investigational drugs;
11. Unwillingness or inability to provide written informed consent;
12. Other contraindications to study treatment;
13. Psychiatric disorders or cognitive impairment limiting legal competency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-07-16 (Estimated); Study Completion 2030-07-16 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
2-Year Progression-Free Survival Rate (PFS) | 2-year
  2-year failure free survival time from the randomization to the first treatment failure or death

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangdong, China

IPD SHARING:
Plan to Share IPD: No